CLINICAL TRIAL: NCT02323061
Title: Brain Computer Interface（BCI） System for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4055037
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BCI-robot (I) (Experimental): EEG guided training based on ipsilesional EEG signals; Training for 20 sessions
  Interventions: Procedure: BCI using EEG signals
- BCI-robot (IC) (Experimental): EEG guided training based on both ipsilesional and contralesional EEG signals; Training for 20 sessions
  Interventions: Procedure: BCI using EEG signals
- robot (Placebo Comparator): Training for 20 sessions
  Interventions: Procedure: BCI using EEG signals

INTERVENTIONS:
Procedure: BCI using EEG signals — A robot hand will be used and controlled by the system in real time based on EEG pattern for identification of motion intention for hand movements in the cortex.

SUMMARY:
A BCI system for stroke subjects will be designed in an attempt to train the motor-related areas in their brains responsible for hand open/close function. A robot hand will be used and controlled by the system in real time based on EEG pattern for identification of motion intention for hand movements in the motor cortex. A randomized controlled trial study design will be adopted. All subjects will be assessed by clinical assessments including FMA and neuroimaging assessments using multimodal MR techniques before and after the training to evaluate training effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Sufficient cognition to follow simple instructions, as well as understand the content and purpose of the experiment;
2. Subcortical ischemic lesion within the territory of the middle cerebral artery;
3. Have moderate to severe motor disability at the paretic upper limb (assessed by Fugl-Meter Assessment (FMA), Modified Ashworth Score of fingers (MAS), and Action Research Arm Test(ARAT)).
4. Hemiparesis resulting from a single unilateral lesion of the brain with onset at least 6 months before data collection.

Exclusion Criteria:

1. Severe hand spasticity, open hand wound or hand deformity;
2. Visual field deficits;
3. Aphasia, neglect, and apraxia,
4. Participation in any therapeutic treatment ("outside therapy") performed with the paralyzed arm during the planned study - including baseline and follow up.
5. History of alcohol, drug abuse or epilepsy,
6. Bilateral infracts,
7. Uncontrolled medical problems,
8. Serious cognitive deficits,
9. Other MRI contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
FMA-UE | 6-month followup
ARAT | 6-month followup

SECONDARY OUTCOMES:
MAS | 6-month followup
MRI | 6-month followup

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lau CCY, Yuan K, Wong PCM, Chu WCW, Leung TW, Wong WW, Tong RKY. Modulation of Functional Connectivity and Low-Frequency Fluctuations After Brain-Computer Interface-Guided Robot Hand Training in Chronic Stroke: A 6-Month Follow-Up Study. Front Hum Neurosci. 2021 Jan 20;14:611064. doi: 10.3389/fnhum.2020.611064. eCollection 2020. PMID 33551777
- [Derived] Yuan K, Wang X, Chen C, Lau CC, Chu WC, Tong RK. Interhemispheric Functional Reorganization and its Structural Base After BCI-Guided Upper-Limb Training in Chronic Stroke. IEEE Trans Neural Syst Rehabil Eng. 2020 Nov;28(11):2525-2536. doi: 10.1109/TNSRE.2020.3027955. Epub 2020 Nov 6. PMID 32997632